CLINICAL TRIAL: NCT02541058
Title: Non-Invasive Chromosomal Evaluation of 22q11.2 Using Cell-free Fetal DNA From Maternal Plasma
Brief Title: Non-Invasive Chromosomal Evaluation of 22q11.2
Acronym: 22Q
Status: Completed | Type: Observational
Sponsor: Cindy Cisneros (Industry)
Responsible Party: Sponsor-Investigator, Cindy Cisneros, CRA, Roche Sequencing Solutions
Organization: Roche Sequencing Solutions (Industry)
Other Study IDs: AD202
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: 22q.11.2 Deletion/Duplication
Keywords: Velocardiofacial Syndrome; Shprintzen Syndrome; Conotruncal Defects; Chromosomal Abnormalities; 22q, 22q.11.2; deletion; duplication
MeSH Terms: conditions — DiGeorge Syndrome; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Confirmed 22q.11.2 deletion/duplication
- Suspected 22q.11.2 deletion/duplication

SUMMARY:
This study is being conducted to develop and evaluate a cell-free fetal DNA test (Harmony) for non-invasive prenatal detection of 22q11.2 chromosomal deletion or duplication.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age and able to provide consent or, if under the age of 18, the patient has parental consent and child assent provided as required by the governing ethics committee.
2. If pregnant, patients must have a singleton pregnancy and be at least 10 weeks gestation at the time of the study blood draw.
3. Patients must meet at least one of the following conditions at the time of enrollment:

   1. are pregnant with abnormal fetal cardiac findings on ultrasound and is undergoing evaluation with prenatal genetic testing or planned post-natal genetic testing in the immediate newborn period;
   2. are pregnant with fetal ultrasound findings consistent with a 22q11.2 deletion/duplication phenotype and is undergoing evaluation with prenatal genetic testing or planned post-natal genetic testing in the immediate newborn period;
   3. are pregnant with a fetus known to have a 22q11.2 deletion/duplication confirmed by genetic testing with documentation is available;
   4. are biologically related parent of an enrolled child has chromosomal deletion/duplication in the region of 22q11.2;
4. If the site is selected to enroll control patients, they must be pregnant women undergoing prenatal genetic evaluation for 22q11.2 deletion/duplication.

Exclusion Criteria

Patients meeting any of the following criteria will be excluded from the study:

1. Patient has history of malignancy treated with chemotherapy and/or major surgery, or bone marrow transplant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women carrying a fetus at risk or a confirmed fetus with 22q11.2 deletion/duplication. A person confirmed to have 22q11.2 deletion/duplication or a biologically related parent of a child that has chromosomal deletion/duplication in the region of 22q11.2.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2015-06; Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Performance of Ariosa 22q.11.2 deletion/duplication assay in prenatal patients | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ong, MD, Study Director — Roche Sequencing Solutions
Locations (1):
- The Fetal Medicine Foundation Belgium, Brussles, Belgium

IPD SHARING:
Plan to Share IPD: Undecided